CLINICAL TRIAL: NCT06493929
Title: Mechanical Power As a Predictor for Weaning in Chronic Obstructive Pulmonary Disease Patients :Prospective Cohort Study.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Moustafa, Assistant Lecturer, Assiut University
Other Study IDs: Mechanical Power
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-07

CONDITIONS: Mechanical Power
Keywords: Mechanical power; Weaning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Paients with Successful weaning from Mechanical Ventilation: The criteria for successful extubation: successful extubation was defined as the ability to maintain spontaneous breathing for at least 48 h, without any ventilatory support.
  Interventions: Other: Chest ultrasound; Other: Calculation of Mechanical Power on the first day of intubation and before First trial of weaning:
- Patients with failed weaning from Mechanical Ventilation: failure extubation was defined as the reconnection to ventilator (invasive or noninvasive) within 48 h due to respiratory failure or other reasons. Extubation and the reconnection to ventilator were all based on SBT results and physicians' decision (5,9).

INTERVENTIONS:
Other: Chest ultrasound — to assess diaphragmatic excursion (DE(. M-mode was used to record the movement of the diaphragm during tidal breathing when the sampling line and diaphragm were as vertical as possible (not < 70°). The data was measured from the first respiratory cycle at 0 min after SBT.
  Groups: Paients with Successful weaning from Mechanical Ventilation
Other: Calculation of Mechanical Power on the first day of intubation and before First trial of weaning: — Total respiratory rate (RR). Positive end-expiratory pressure (PEEP) (the external or applied PEEP) recorded, not the total PEEP, or intrinsic PEEP. The plateau pressure (Pplat) was measured during an inspiratory pause on the ventilator. Peak inspiratory pressure (Ppeak) should be obtained while the patient is relaxed, not coughing or moving in bed. MP was calculated according to Gattinoni's simplified mechanical power equation as follows (3,8):
  MP(J/min)=0.098×VT×RR×(Ppeak-0.5×ΔP).
  Groups: Paients with Successful weaning from Mechanical Ventilation

SUMMARY:
The primary objective is to evaluate the mechanical power as a predictor of weaning of mechanical ventilation in COPD patients hospitalized in the respiratory intensive care unit of Assiut University Hospital The secondary objective is to compare between mechanical power and diaphragmatic excursion (DE) assessed by ultrasound as a predictor of weaning in these patients. Also, to investigate the association between MP and DE and mortality in these patients

DETAILED DESCRIPTION:
Acute exacerbation of chronic obstructive pulmonary disease (AECOPD), a public health problem that is characterized by persistent airflow limitation ,it develops when there is a significant exposure of irritants causing an inflammatory response in the lungs, it is a common cause of respiratory failure which require hospital admission that is associated with increased medical costs.

The World Health Organization reported that COPD was the fifth most common disease globally in 2020, with a prevalence of 7.8-19.7% in adults. Approximately, 60% of patients with COPD admitted with hypercapnic respiratory failure.

Acute exacerbations of chronic obstructive pulmonary disease (COPD) is characterized by acute worsening of respiratory symptoms associated with the development of severe airflow limitation, gas trapping, dynamic hyperinflation and intrinsic positive end-expiratory pressure (PEEPi). In the most severe cases, these exacerbations may cause acute respiratory failure, which may require mechanical ventilation.

The process of weaning from mechanical ventilation remains one of the most critical challenges in patients underwent mechanical ventilation in the intensive care unit (ICU). The multidisciplinary team must study the optimal time for weaning from the mechanical ventilator as premature weaning may lead to weaning failure and thus increase the risk of hospital acquired infections, costs of care, length of ICU stay, Morbidity and Mortality.

Current guidelines recommend several indices applied at the bedside to predict successful weaning from mechanical ventilation. A spontaneous breathing trial (SBT) is an appropriate way to prepare the patient for extubation; however, even after successful SBT, failure rates and subsequent reintubation can exceed 20% in the highest-risk patient.

Mechanical power (MP) is the energy delivered by the ventilator to the entire respiratory system per time unit and combines all factors affecting the energy load of the respiratory system, including pressure, tidal volume, flow rate and respiratory rate.

MP is primarily calculated as the product of the applied airway pressure and minute ventilation and can be used as an estimate of the workload exerted on the respiratory muscles during spontaneous breathing.

MP is a major determinant to ensure adequate gas exchange in the body and a key factor in assessing the ability of a patient to successfully wean from mechanical ventilation.

Therefore, a larger scale clinical study is needed to further verify the relationship between MP and weaning outcomes in all critically ill mechanically ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* All COPD mechanically ventilated patients admitted to respiratory intensive care unit and eligible for weaning according to European respiratory society 2016 (5).

Exclusion Criteria:

- 1. Patients with associated lung pathology that may alter lung mechanics (Bronchiectasis, interstitial lung diseases, lung scarring) will be excluded from the study.

2. Tracheostomized patients.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients who are mechanically ventilated in Respiratory ICU in Assiut University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
1. Evaluation the efficacy of MP as a predictor of weaning for COPD patients. | 2 years
  Evaluation the efficacy of MP as a predictor of weaning for COPD patients.

SECONDARY OUTCOMES:
1-MP as a predictor of patient's mortality. | 2 years
  MP as a predictor of patient's mortality.
2-MP and duration of hospital stay and ICU stay. | 2 years
  MP and duration of hospital stay and ICU stay.
3-MP and ventilator induced lung injury. | 2 years
  THE ASSOCIATION BETWEEN VALUE OF MP and ventilator induced lung injury.
4-Correlation analysis between mechanical power and other parameters of weaning: Respiratory rate, Rapid shallow breathing index, Heart Rate and Expiratory Tidal volume in evaluation of prognosis in COPD patients. | 2 years
  Correlation analysis between mechanical power and other parameters of weaning: Respiratory rate, Rapid shallow breathing index, Heart Rate and Expiratory Tidal volume in evaluation of prognosis in COPD patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu J, Lee MR, Chen CT, Lin YT, How CK. Predictors of Successful Weaning from Noninvasive Ventilation in Patients with Acute Exacerbation of Chronic Obstructive Pulmonary Disease: A Single-Center Retrospective Cohort Study. Lung. 2021 Oct;199(5):457-466. doi: 10.1007/s00408-021-00469-z. Epub 2021 Aug 21. PMID 34420091
- [Background] Mohamed-Hussein AAR, Makhlouf HA, Selim ZI, Gamaleldin Saleh W. Association between hand grip strength with weaning and intensive care outcomes in COPD patients: A pilot study. Clin Respir J. 2018 Oct;12(10):2475-2479. doi: 10.1111/crj.12921. Epub 2018 Sep 23. PMID 29931773
- [Background] Yan Y, Xie Y, Chen X, Sun Y, Du Z, Wang Y, Li X. Mechanical power is associated with weaning outcome in critically ill mechanically ventilated patients. Sci Rep. 2022 Nov 16;12(1):19634. doi: 10.1038/s41598-022-21609-2. PMID 36385129
- [Background] Azizi BA, Munoz-Acuna R, Suleiman A, Ahrens E, Redaelli S, Tartler TM, Chen G, Jung B, Talmor D, Baedorf-Kassis EN, Schaefer MS. Mechanical power and 30-day mortality in mechanically ventilated, critically ill patients with and without Coronavirus Disease-2019: a hospital registry study. J Intensive Care. 2023 Apr 6;11(1):14. doi: 10.1186/s40560-023-00662-7. PMID 37024938
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Background] Leonov Y, Kisil I, Perlov A, Stoichev V, Ginzburg Y, Nazarenko A, Gimelfarb Y. Predictors of successful weaning in patients requiring extremely prolonged mechanical ventilation. Adv Respir Med. 2020;88(6):477-484. doi: 10.5603/ARM.a2020.0151. PMID 33393639
- [Background] Zhang X, Yuan J, Zhan Y, Wu J, Liu B, Zhang P, Yu T, Wang Z, Jiang X, Lu W. Evaluation of diaphragm ultrasound in predicting extubation outcome in mechanically ventilated patients with COPD. Ir J Med Sci. 2020 May;189(2):661-668. doi: 10.1007/s11845-019-02117-1. Epub 2019 Nov 6. PMID 31691888
- [Background] Paudel R, Trinkle CA, Waters CM, Robinson LE, Cassity E, Sturgill JL, Broaddus R, Morris PE. Mechanical Power: A New Concept in Mechanical Ventilation. Am J Med Sci. 2021 Dec;362(6):537-545. doi: 10.1016/j.amjms.2021.09.004. Epub 2021 Sep 28. PMID 34597688
- [Background] Akella P, Voigt LP, Chawla S. To Wean or Not to Wean: A Practical Patient Focused Guide to Ventilator Weaning. J Intensive Care Med. 2022 Nov;37(11):1417-1425. doi: 10.1177/08850666221095436. Epub 2022 Jul 11. PMID 35815895